CLINICAL TRIAL: NCT01996384
Title: Acupuncture Augmentation of Lidocaine for the Treatment of Provoked, Localized vulvodynia-a Feasibility and Acceptability Pilot Study
Brief Title: Provoked, Localized Vulvodynia Treatment With Acupuncture and Lidocaine Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon College of Oriental Medicine (Other)
Collaborators: National Vulvodynia Association (Other); Council of Colleges of Acupuncture and Oriental Medicine (Unknown); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lee Hullender Rubin, DAOM, LAc, Adjunct Research Faculty, Oregon College of Oriental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 9664
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Provoked, Localized Vulvodynia; Provoked Vestibulodynia; Vulvar Vestibulitis; Vulvodynia
Keywords: Vulvodynia; Provoked, localized vulvodynia; vulvar vestibulitis; provoked vestibulodynia; vulvovaginal pain; vulvar pain; vaginal pain; chronic pain; lidocaine; numbing agent; anesthetic cream; acupuncture; electroacupuncture; electrical stimulated acupuncture; manual acupuncture; classical acupuncture; non-classical acupuncture; Traditional Chinese Medicine; TCM; Chinese medicine; Acupuncture and Oriental Medicine; AOM; treatment; feasibility; pilot study; Patient Reported Outcomes Measure Information System; Tampon Test; cotton swab test; pain diary; Research Electronic Data Capture; REDCap
MeSH Terms: conditions — Vulvar Vestibulitis; Vulvodynia; Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classical Acupuncture + Lidocaine (Experimental): Study participants will attend 18 classical acupuncture sessions, twice a week for Weeks 1-6, and once a week for Weeks 7-12. A standardized acupuncture treatment will be assigned with classical acupuncture points and may or may not be stimulated with electroacupuncture. Very thin needles (0.18mm) will be inserted into locations either on the front or the back of the body and may be placed near or far from the affected area based on up to three Traditional Chinese Medicine Diagnosis categories. Study participants will also be asked to gently apply 5% lidocaine cream four times daily (breakfast, lunch, dinner, and before bed).
  Interventions: Procedure: Classical Acupuncture; Drug: Lidocaine
- Non-classical acupuncture + lidocaine (Active Comparator): Study participants will attend 18 non-classical acupuncture sessions, twice a week for Weeks 1-6, and once a week for Weeks 7-12. A standardized acupuncture treatment will be assigned with non-classical acupuncture points and may or may not be stimulated with electroacupuncture. Very thin needles (0.18mm) will be inserted into locations either on the front or the back of the body and may be placed near or far from the affected area. Study participants will also be asked to gently apply 5% lidocaine cream four times daily (breakfast, lunch, dinner, and before bed).
  Interventions: Procedure: Non-classical acupuncture; Drug: Lidocaine

INTERVENTIONS:
Procedure: Classical Acupuncture — Very thin needles (0.18mm) will be inserted into locations either on the front or the back of the body and may be placed near or far from the affected area. No needles will be inserted into the genital region. Locations needled will be in classical acupuncture points. On even-numbered visits, the needles may be electrically stimulated via an electro-acupuncture machine. Needles will be retained for 30 minutes per study visit. Acupuncture needles used are 0.18x30-40mm, manufactured by Dong Bae Corporation (DBC), Korea. The electrical acupuncture device is Pantheon Research Electrical Stimulator 8c, United States.
  Arms: Classical Acupuncture + Lidocaine
Procedure: Non-classical acupuncture — Very thin needles (0.18mm) will be inserted into locations either on the front or the back of the body and may be placed near or far from the affected area. No needles will be inserted into the genital region. Locations needled will be in non-classical acupuncture points. On even-numbered visits, the needles may be electrically stimulated via an electro-acupuncture machine. Needles will be retained for 30 minutes per study visit. Acupuncture needles used are DBC Brand, Korea, 0.18x30-40mm. The electrical acupuncture device is Pantheon Research Electrical Stimulator 8c, United States.
  Arms: Non-classical acupuncture + lidocaine
Drug: Lidocaine — Study participants will gently apply 5% lidocaine cream four times daily to vulvar area.
  Other Names: 5% Lidocaine cream

SUMMARY:
The investigators research project is a randomized, controlled, single-blinded, feasibility pilot study. The investigators will study the feasibility of a novel treatment for women with Provoked Localized Vulvodynia (PLV) with acupuncture and 5% lidocaine cream. Lidocaine is a numbing agent and common first treatment for this disorder. Acupuncture is a treatment commonly used for other pain disorders. The investigators will compare two types of acupuncture (classical and non-classical) as a treatment for PLV, in addition to 5% lidocaine cream. Researchers want to determine if acupuncture is acceptable and convenient to women with PLV. The investigators hypothesize that classical acupuncture and 5% lidocaine cream will be better than non-classical acupuncture and 5% lidocaine cream to decrease PLV pain.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blinded, pilot trial to study the feasibility and acceptability of acupuncture and 5% lidocaine. Patients will be recruited from the patient population of the Oregon Health & Science University Vulvar Health Clinic. Thirty (30) patients with PLV will be enrolled as study participants into the study. Fifteen (15) will be allocated in the treatment (classical) acupuncture + 5% lidocaine group and fifteen (15) will be allocated in the control (non-classical) acupuncture + 5% lidocaine group via a computer generated randomization program to balance allocation based on four variables: pain intensity, smoking status, body mass index, and pain duration.

The acupuncturist will interview each patient and perform an exam of the pulse and tongue. A standardized acupuncture treatment will be assigned, and both groups will receive 18 acupuncture treatments that follow a standardized protocol on classical or non-classical acupuncture points, with or without mild electrical stimulation. All study participants will self-apply lidocaine cream to their genital region four times daily during the study.

ELIGIBILITY:
Inclusion Criteria:

* Literate, English speaking, premenopausal, women meeting Friedrich's criteria for Provoked, localized vulvodynia
* Reported introital dyspareunia longer than three months duration;
* Average pain score greater than 4 on Visual Analog Scale (VAS) at enrollment with cotton swab test and Tampon Test;
* Able to insert an Original Regular Tampax™ tampon.

Exclusion Criteria:

* Co-existing conditions leading to dyspareunia including generalized unprovoked vulvodynia, atrophic vaginitis, vulvovaginal dermatoses (e.g. lichen sclerosus), or genital infection (e.g. herpes simplex virus or yeast infection).
* Pregnant or postpartum and breastfeeding;
* Use of neuromodulator medications (e.g. Serotonin Norepinephrine Reuptake Inhibitors (SNRIs), Tricyclic Antidepressants, or anti-seizure medications) started in the last six months. If taken for longer, must be on a stable dose for at least six months and still report moderate to severe pain. Selective Serotonin Reuptake Inhibitors (SSRIs) are allowed;
* Postmenopausal as defined by surgical or natural menopause (no menses for 12 months);
* Chronic pelvic pain defined as daily, non-menstrual pain in pelvis or lower abdomen for longer than three months duration;
* Must be able to refrain from other treatments for PLV including non-traditional options (e.g. other medications, physical therapy, sex therapy, acupuncture, naturopathic remedies) during the course of the study (6 months).
* Use of SNRIs, lidocaine, or acupuncture within the last three months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tampon Test | Weeks 1 and 12 study period
  Primary outcome variable will be to measure the change in the reported pain of the "Tampon Test" (mean at Week 1) to the reported pain of "Tampon Test" (mean of Week 12);
  Every week, study participants will be asked to fully insert and remove a tampon and rate the level of pain with insertion on a 10-point Visual Analog Scale (0 indicating no pain, 10 indication worst possible pain).

SECONDARY OUTCOMES:
Cotton Swab test | Weeks -4, -3, -2, -1, 0, 1, 12 or 13 and 24.
  Secondary outcome variable will compare the "Cotton Swab Test" with a blinded assessor reported pain at three timepoints. 1) change in reported pain at (mean at Weeks -2, -1, 0, and 1) to the reported pain (mean at Weeks 12 and 13; 2) change in reported pain (means Weeks -2, -1, 0, and 1) to the reported pain (mean at Week 24); 3) change in reported pain (mean at Week 12) to (mean at Week 24).
  Vestibular tenderness will be assessed by light touch with a cotton swab by a blinded assessor to the study participant's: 1) vestibule (cotton swab test) at four defined points (1:00, 5:00, 7:00, and 11:00); 2) the perineum; 3) labia majora (2:00 and 8:00), and 4) labia minora (4:00 and 10:00). Tenderness at each location will be rated by the Study Participant on a 10-point scale (0 indicating no pain, 10 indicating worst possible pain).
Patient Reported Outcomes Measurement Information System (PROMIS) Scales | At baseline visit, 6 weeks, 12 weeks, and 24 weeks
  Assess changes in scores quality of life, vaginal discomfort, pain intensity, pain interference and behavior, anxiety, and depression at 6 weeks, 12 weeks, and 24 weeks compared to baseline.
Satisfaction | Weeks 12 and 24
  Using 5-point scales (Very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, Very dissatisfied), Study participants will be asked how satisfied they are with the study interventions and how satisfied they are with their pain relief.
Expectation | Week 1
  Study participants will be asked about how much they 'expect' the study interventions will or will not help, how much they 'think' the intervention will or will not help, and how much they 'feel' about the intervention will or will not help via 10-point scales.
Feasibility | Weeks 12 and 24
  Assess feasibility by the number of study participants enrolled.
Acceptability | Weeks 12 and 24
  Assess acceptability by the number of study visits attended by participants enrolled.
Tampon Test | Weeks 1 and 6; Weeks 1 and 24
  Secondary outcome variables will be to:
  1. measure the change in reported pain of the "Tampon Test" (mean at Week 1) to the reported pain of "Tampon Test" (mean of Week 6);
  2. measure the change in reported pain of the "Tampon Test" (mean at Week 1) to the reported pain of "Tampon Test" (mean of Week 24);
  3. measure the change in reported pain of the "Tampon Test" (mean at Week 12) to the reported pain of "Tampon Test" (mean of Week 24).
  Every week, study participants will be asked to fully insert and remove a tampon and rate the level of pain with insertion on a 10-point Visual Analog Scale (0 indicating no pain, 10 indication worst possible pain).

OTHER OUTCOMES:
Traditional Chinese Medicine (TCM) Diagnosis Category | Week 1
  TCM Diagnosis Category will be recorded and tracked by the primary investigator to determine if it may be a potential predictor of treatment response.
24-hour mean pain score | Baseline, Weeks 6, 12, and 24
  In a daily pain diary, study participants will be asked to record the level of pain they are experiencing based via the 10-point VAS scale (0 indicates no pain, 10 indicates worst possible pain).
Frequency of intercourse | Baseline, Weeks 6, 12, and 24
  In a daily pain diary, study participants will be asked to record if they engaged in intercourse within the last 24 hours.
Intensity of Intercourse pain | Baseline, Weeks 6, 12, and 24
  In a daily pain diary, study participants will be asked to record the level of pain they are experienced with intercourse based via the 10-point VAS scale (0 indicates no pain, 10 indicates worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Lee E Hullender Rubin, DAOM, Principal Investigator — Oregon College of Oriental Medicine
Locations (1):
- Women's Health Research Unit; Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Hullender Rubin LE, Mist SD, Schnyer RN, Chao MT, Leclair CM. Acupuncture Augmentation of Lidocaine for Provoked, Localized Vulvodynia: A Feasibility and Acceptability Study. J Low Genit Tract Dis. 2019 Oct;23(4):279-286. doi: 10.1097/LGT.0000000000000489. PMID 31592976
- See also: Related Info — http://journals.lww.com/jlgtd/Citation/2017/10001/Abstracts.1.aspx